CLINICAL TRIAL: NCT02314676
Title: Phase IV Clinical Study of Pegylated Somatropin (PEG Somatropin) to Treat Growth Hormone Deficiency Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GenSci 004 CT
Record Dates: First submitted 2014-11-27; First posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Dwarfism, Pituitary
MeSH Terms: conditions — Dwarfism, Pituitary

ARMS (1):
- PEG-somatropin (Experimental)
  Interventions: Biological: PEG-somatropin

INTERVENTIONS:
Biological: PEG-somatropin

SUMMARY:
This study evaluates the safety and efficiency of Pegylated Somatropin (PEG Somatropin) Injection in the treatment of endogenous growth hormone deficiency (GHD) in the broad population of children. Half of participants will receive the high dose, while the other half will receive the low dose.

ELIGIBILITY:
Inclusion Criteria:

* Before starting treatment, according to the medical history, clinical symptoms and signs, GH stimulation test and imaging examination, patients are diagnosed as GHD.
* According to the height statistical data of Chinese children's physique development in nine cities in 2005, height is lower than the third percentile of growth curve of normal children with the same age and gender.
* Height velocity (HV) ≤5.0 cm/yr.
* GH stimulation test with two different mechanisms affirms that GH peak concentration of patients' plasma <10.0ng/ml.
* Bone age (BA) ≤9 years in girls and ≤10 years in boys, at least 1 year less than his/her chronological age (CA).
* Be in preadolescence (Tanner stage 1) and have a CA ≧ 3 years.
* Receive no prior GH treatment within 6 months.
* Sign informed consent.

Exclusion Criteria:

* People with abnormal liver or kidney function (ALT> 2 times the upper limit of normal value, Cr> the upper limit of normal value).
* Patients positive for hepatitis B core antigen (HBc), hepatitis B surface antigen (HBsAg) or hepatitis B e antigen (HBeAg).
* People with known highly allergic constitution or allergy to the drug of the study.
* People with severe cardiopulmonary, hematological and malignant tumors diseases or general infection and immune deficiency.
* Potential tumor patients (family history).
* Diabetic.
* Abnormal growth and development, such as Turner syndrome, constitutional delay of growth and puberty, Laron syndrome, growth hormone receptor deficiency, girls of growth retardation without excluding abnormal chromosome.
* Subjects took part in other clinical trial study within 3 months.
* Other conditions which in the opinion of the investigator preclude enrollment into the study.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Actual height of the patient after treatment compared with the mean height of the population and the standard deviation (SD) of the height of the population for that chronological age | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Junfen Fu, Ph.D, Principal Investigator — Children's Hospital Affiliated to Medical College of Zhejiang University
Locations (2):
- China (2):
  - First People's Hospital of Wuhu, Wuhu, Anhui
  - Children's Hospital Affiliated to Zhejiang University, Hangzhou, Zhejiang